CLINICAL TRIAL: NCT01691469
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover, Oral Bioequivalence Study in Healthy, Adult, Human Subjects Under Fed Conditions.
Brief Title: Bioequivalence Study of Montelukast Sodium Oral Granules 4mg Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 540-10
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Montelukast Sodium; crossover
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast Sodium Oral Granules (Experimental): Montelukast Sodium Oral Granules 4mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Montelukast sodium
- SINGULAIR (Active Comparator): (Montelukast sodium) Oral Granules 4mg of Merck Sharp & Dohme Ltd., USA
  Interventions: Drug: Montelukast sodium

INTERVENTIONS:
Drug: Montelukast sodium — Montelukast Sodium Oral Granules 4mg
  Other Names: SINGULAIR

SUMMARY:
This is an open label, randomised, balanced, two-treatment, two-period, two-sequence, single dose, crossover, oral bioequivalence study.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover, oral bioequivalence study of Montelukast Sodium Oral Granules 4mg of Dr. Reddy's Laboratories Limited, India comparing with that of SINGULAIR® (Montelukast sodium) 4mg oral granules of Merck Sharp & Dohme Ltd., USA in healthy, adult, human subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill the following criteria to be considered for inclusion into this study.

* Healthy subjects within the age range of 18 to 50 years.
* A body mass index between 18.5 to 24.9 Kg/m2
* Given written informed consent to participate in the study.
* Absence of disease markers of HIV 1 & 2, hepatitis B & C virus and RPR.
* Absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history and physical examination during the screening.
* A normal 12-lead ECG.
* A normal chest X-ray (PA view).
* Compliance with the requirement of the entire protocol.
* No history or no evidence of hypersensitivity to Montelukast and to any component of the formulation.
* No history of gastrointestinal problems (ulcers).
* No history of significant systemic diseases.
* No history of psychiatric disorders.
* No history of allergic rash.
* No history of addiction to any recreational drug or drug dependence.
* No donation of blood (one unit or 350 mL) within 90 days prior to study check in.
* No Participation in any clinical study within the past 90 days.
* No receipt of any prescription drugs or over-the-counter drugs (e.g.: Cold preparations, and antacid preparations vitamins and natural products used for therapeutic benefits), within two weeks prior to study check-in.
* No history of dehydration from dialThea, vomiting or any other reason within a period of24.0 hours prior to study check-in.
* No family history of neurological disorders. Not consumed alcohol and xanthine containing food and beverages (chocolates, tea, coffee or cola drink:s), cigarettes and tobacco products, for at least 48.0 hours prior to study check-in.
* Negative results for drugs of abuse (Benzodiazepines, Cocaines, Opioids, Amphetamines, Ca1U1abinoids and Barbiturates) in urine during the day of study check-in.
* Not consumed grapefruit (mosumbi/sweet lime) juice within the 48.0 hours prior to study check-in.
* Negative alcohol breath analysis during the study check-in.
* Female volunteers demonstrating a negative pregnancy test.
* If study volunteer is a female volunteer and is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.

or is postmenopausal for at least 1 year. or is surgically . sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy has been performed on the study volunteer).

Exclusion Criteria The subjects were excluded based on the following criteria.

* History of seizures.
* Received pharmacological agents known to significantly induce or inhibit drug metabolizing enzymes within 14 days of the start of the study.
* History of alcohol consumption for more than two units/day (1 unit = 30 mL of spirit/or 1 pint of beer), or having consumed alcohol within 48 hours prior to check-in.
* High caffeine (more than 5 cups of coffee or tea/day) or tobacco (more than 9 cigarettes/beedies/cigars per day) consumption.
* History of difficulty with donating blood or difficulty in accessibility of veins.
* An unusual or abnormal diet, for whatever reason e.g. because of fasting due to religious reasons.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Area under curve(AUC) | Pre-dose (0.00) and 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 7.50, 8.00, 8.50, 9.00, 12.00, 16.00, 20.00 and 24.00 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: A. Jayachandra Reddy, Dr., Principal Investigator — Axis Clinicals Limited
Locations (1):
- AXIS Clinicals Limited,, Hyderabad, Andhra Pradesh, India